CLINICAL TRIAL: NCT06580925
Title: Effects of Dynamic Taping on Shoulder Strength, Fatigue, Corticomotor Control and Neuromuscular Control
Brief Title: Effects of Dynamic Taping on Shoulder Isokinetics Strength and Muscle Fatigue.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yin-Liang Lin, Associate Professor, National Yang Ming Chiao Tung University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NYCU112007AF-1
Record Dates: First submitted 2024-08-27; First posted 2024-08-30 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Dynamic Tape; Kinesio Taping; Strength; Fatigue
MeSH Terms: conditions — Fatigue | interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- sham tape (Sham Comparator)
  Interventions: Device: sham tape
- kinesio tape (Active Comparator)
  Interventions: Device: kinesio tape
- dynamic tape (Experimental)
  Interventions: Device: dynamic tape

INTERVENTIONS:
Device: sham tape — sham
  Arms: sham tape
Device: kinesio tape — Kinesio taping will be applied to correct shoulder posture and facilitate shoulder external rotators
  Arms: kinesio tape
Device: dynamic tape — Dynamic tape will be applied to correct shoulder alignment and assist concentric contraction and eccentric control of external rotators
  Arms: dynamic tape

SUMMARY:
Maintaining shoulder stability requires good neuromuscular control. Imbalances in shoulder internal and external rotator strength may increase the risk of shoulder injuries in overhead athletes, and the compromised fatigue resistance of the external rotators may worsen this imbalance during sports activities. Additionally, poor scapular neuromuscular control is associated with shoulder problems, such as shoulder impingement syndrome. Previous research has shown that individuals with shoulder impingement syndrome exhibit poor scapular motion control and altered corticomotor control. Poor scapular motion control, pain, functional impairment, and changes in corticomotor control interact to form a vicious cycle. Various treatments have been attempted to improve neuromuscular control, including taping. Most past studies have focused on the efficacy of rigid tape and kinesio tape, while dynamic tape has gained popularity in recent years. Due to its material properties, dynamic tape is theoretically able to absorb loads, provide force, and correct movements. However, there is currently a lack of evidence supporting the effectiveness of dynamic tape. No research has yet explored whether dynamic tape can provide force to increase muscle strength and reduce fatigue or whether its movement correction functions can improve neuromuscular control and corticomotor control. Therefore, this project plans to conduct an experiment to investigate the effects of dynamic tape on external rotator strength and fatigue in recreational overhead athletes, as well as its impact on neuromuscular control and corticomotor excitability in recreational overhead athletes with shoulder impingement syndrome. In the experiment, 37 healthy recreational overhead athletes will participate in three testing sessions spaced one week apart, receiving kinesio tape, dynamic tape, and sham tape. After taping, they will perform fatigue-inducing activities. Isokinetic strength of internal and external rotators will be measured before taping, after taping, and after fatigue-inducing activities to observe the effects of dynamic tape on muscle strength and fatigue compared to kinesio tape and sham tape.

ELIGIBILITY:
Inclusion Criteria:

* practice overhead exercise more than six hours a week
* aged 18 to 40 years old

Exclusion Criteria:

* have a history of dislocation, fracture, or surgery of neck or upper extremity
* a history of pain or injuries over the neck or upper extremities within the past 12 months
* brain injury and neurological impairment
* arm elevation angle is less than 150 degrees

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-03-24 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Shoulder isokinetic muscle strength | Change from baseline shoulder isokinetic muscle strength after application of taping (about 4 minutes) and execution of a fatigue protocol (about 5 minutes)
  Shoulder isokinetic internal and external muscle strength will be measured by dynamometer in 2 modes (concentric/concentric, concentric/eccentric) at 2 angular velocities (60°/s & 240°/s), 1 set of 5 repetitions for each angular velocities. Shoulder isokinetic muscle strength will be normalized by body weight (BW) and described with peak torque/BW (N·m·kg-1).

SECONDARY OUTCOMES:
Median frequency | Change from baseline shoulder isokinetic muscle strength after execution of a fatigue protocol (about 5 minutes)
  The median frequency calculated from electromyographic data of shoulder internal and external rotators. The percentage change in median frequency will be calculated and will be described with percentage (%)

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taipei city, Taiwan